CLINICAL TRIAL: NCT01160133
Title: To Evaluate the Physical Effects of Systane(R) Lubricant Eye Drops Compared to Refresh Tears(R) Lubricant Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMA-09-67
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Systane; Refresh Tears; Dry Eye; Moderate to Severe Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane (Experimental): Systane Lubricant Eye Drops
  Interventions: Other: Systane
- Refresh Tears (Experimental): Refresh Tears Lubricant Eye Drops
  Interventions: Other: Refresh Tears

INTERVENTIONS:
Other: Systane — Systane Lubricant Eye Drops (1-2 drops in each eye, four times per day)
  Arms: Systane
Other: Refresh Tears — Refresh Tears Lubricant Eye Drops (1-2 drops in each eye, four times per day)
  Arms: Refresh Tears

SUMMARY:
This is a multi-site, randomized, investigator-masked study to evaluate the physical effects of Systane(R) versus Refresh Tears(R) in subjects with moderate to severe dry eye. It is a 6-week, perspective, randomized, active-controlled, investigator-masked, parallel group study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older of any sex and any race, with a score of at least 2 (some of the time) on the subject-assessed Symptom Eligibility question.
* A sodium fluorescein corneal staining sum of ≥ 3 in either eye.
* A best-corrected visual acuity of 0.6 logMAR or better in each eye as assessed using an ETDRS chart.

Exclusion Criteria:

* A history or evidence of ocular or intraocular surgery in either eye within the past 6 months.
* Lasik patients can be included if lasik surgery was greater than 6 months prior to the initiation of the study.
* A history of intolerance or hypersensitivity to any component of the study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate physical effects of Systane and Refresh Tears in subjects to moderate to severe dry eye. | Baseline to visit 3 (Day 42)
  This is a descriptive study in which changes from baseline in Tear Break up Time, corneal staining, and the Ocular Symptoms Questionnaire will be evaluated by treatment group at every visit. The outcome of the IDEEL questionnaire at Visit 3 will be compared to Visit 1 by treatment group; the results of treatment satisfaction questionnaires will be tabulated by treatment at Visit 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Vasan Eye Care Hospital, Saidāpet, Channai, India